CLINICAL TRIAL: NCT01710501
Title: A Phase II Randomized, Dose Ranging, Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of Different Doses of MK-5172 When Administered Concomitantly With Peginterferon Alfa-2b and Ribavirin in Treatment Naïve Subjects With Chronic Hepatitis C Virus Infection
Brief Title: A Study of Different Doses of Grazoprevir (MK-5172) Given With Pegylated Interferon Alfa-2b and Ribavirin to Treatment-Naïve Participants With Chronic Hepatitis C (MK-5172-038)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-038; 2012-003333-42 (EudraCT Number)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis C (CHC)
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Grazoprevir 25 mg + PEG-IFN + RBV (Experimental): After a maximum of a 45 day screening window, randomized participants receive 25 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by Response Guided Therapy (RGT). Participants may receive an additional 12 weeks of PEG-IFN plus RBV depending on their Hepatitis C virus ribonucleic acid (HCV RNA) level at Treatment Week (TW) 4.
  Interventions: Drug: Grazoprevir; Biological: pegylated interferon alfa-2b; Drug: Ribavirin; Drug: Placebo
- Grazoprevir 50 mg + PEG-IFN + RBV (Experimental): After a maximum of a 45 day screening window, randomized participants receive 50 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by RGT. Participants may receive an additional 12 weeks of PEG-IFN plus RBV depending on their HCV RNA level at TW 4.
  Interventions: Drug: Grazoprevir; Biological: pegylated interferon alfa-2b; Drug: Ribavirin; Drug: Placebo
- Grazoprevir 100 mg + PEG-IFN + RBV (Experimental): After a maximum of a 45 day screening window, randomized participants receive 100 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by RGT. Participants may receive an additional 12 weeks of PEG-IFN plus RBV depending on their HCV RNA level at TW 4.
  Interventions: Drug: Grazoprevir; Biological: pegylated interferon alfa-2b; Drug: Ribavirin; Drug: Placebo

INTERVENTIONS:
Drug: Grazoprevir — Grazoprevir tablet, orally, once per day at assigned dose
  Other Names: MK-5172
Biological: pegylated interferon alfa-2b — 1.5 mcg/kg/week, administered as a weekly subcutaneous (SC) injection
  Other Names: SCH 054031; PegIntron™; PEG-IFN
Drug: Ribavirin — Ribavirin capsule, orally, twice daily, at a dose of 800 to 1400 mg based on participant weight
  Other Names: Rebetol™; RBV
Drug: Placebo — Placebo to match grazoprevir tablets to maintain dose blinding

SUMMARY:
This is a study designed to compare the safety and efficacy of 3 different doses of grazoprevir (MK-5172) combined with pegylated interferon alfa-2b (PEG-IFN) and ribavirin (RBV) in treatment-naïve participants with genotype 1 (GT1) chronic hepatitis C (CHC). Participants will receive 12 weeks of treatment with grazoprevir combined with Peg-IFN and RBV, and depending on response at Week 4 may go on to receive an additional 12 weeks of treatment with Peg-IFN and RBV.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive
* Chronic, compensated HCV GT1 infection
* Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease, or cirrhosis
* No evidence of cirrhosis or hepatocellular carcinoma by biopsy or noninvasive testing (e.g. FibroScan and/or FibroTest)
* Must agree to use two acceptable methods of birth control from at least 2 weeks prior to first dose and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations

Exclusion Criteria:

* Non-GT1 HCV infection, including a mixed GT infection (with a non-GT1) or a non-typeable genotype.
* Documented to be Human Immunodeficiency Virus (HIV) positive or co-infected with hepatitis B virus
* Hepatocellular carcinoma (HCC) or under evaluation for HCC
* Participating in or has participated in a study with an investigational compound or device within 30 days of signing informed consent
* Diabetic and/or hypertensive with clinically significant ocular examination findings
* Current or history of central nervous system trauma, seizure disorder, stroke or transient ischemic attack
* Chronic pulmonary disease
* Current or history of any clinically significant cardiac abnormalities/dysfunction
* Active clinical gout within the last year
* History of gastric surgery or history of malabsorption disorders
* Active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin)
* Pregnant, lactating, expecting to conceive or donate eggs, or male participant planning to impregnate or provide sperm donation or with a female partner who is pregnant
* Current moderate or severe depression or history of depression associated with hospitalization, electroconvulsive therapy, or severe disruption of daily functions, or suicidal or homicidal ideation and/or attempt, or history of severe psychiatric disorders
* Evidence or history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2013-11-25 (Actual); Study Completion 2014-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lagging M, Brown A, Mantry PS, Ramji A, Weilert F, Vierling JM, Howe A, Gendrano IN 3rd, Hwang P, Zhang B, Wahl J, Robertson M, Mobashery N. Grazoprevir plus peginterferon and ribavirin in treatment-naive patients with hepatitis C virus genotype 1 infection: a randomized trial. J Viral Hepat. 2016 Feb;23(2):80-8. doi: 10.1111/jvh.12464. Epub 2015 Sep 10. PMID 26353843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 136 screened participants, 87 were randomized to treatment at 19 sites worldwide.
Groups:
- Grazoprevir 25 mg + PEG-IFN + RBV: After a maximum of a 45 day screening window, randomized participants received 25 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by RGT. Participants could receive an additional 12 weeks of PEG-IFN plus RBV depending on their HCV RNA level at TW 4.
- Grazoprevir 50 mg + PEG-IFN + RBV: After a maximum of a 45 day screening window, randomized participants received 50 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by RGT. Participants could receive an additional 12 weeks of PEG-IFN plus RBV depending on their HCV RNA level at TW 4.
- Grazoprevir 100 mg + PEG-IFN + RBV: After a maximum of a 45 day screening window, randomized participants received 100 mg grazoprevir in combination with PEG-IFN and RBV for 12 weeks followed by 24 weeks of follow-up as determined by RGT. Participants could receive an additional 12 weeks of PEG-IFN plus RBV depending on their HCV RNA level at TW 4.
Period: Overall Study
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Started | 29 | 28 | 30
Completed | 27 | 28 | 30
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV | Total
Number analyzed (Participants) | 29 | 28 | 30 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (7.9) | 48.5 (12.5) | 46.4 (13.3) | 48.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 18 | 15 | 41
  Male | 21 | 10 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at 12 Weeks After the End of Treatment (SVR12)
Description: Hepatitis C virus ribonucleic acid (HCV RNA) was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. SVR12 was defined as HCV RNA <25 IU/mL (either target detected, unquantifiable or target not detected) 12 weeks after the end of all study therapy.
Time Frame: 12 weeks after end of treatment (up to 36 weeks total)
Population: Participants in the Per-Protocol (PP) Population (all randomized participants receiving ≥1 dose of study treatment and no important protocol deviation) with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 24 | 25 | 26
percentage of participants | 54.2 [32.8 to 74.4] | 84.0 [63.9 to 95.5] | 88.5 [69.8 to 97.6]

2. Primary Outcome: Number of Participants Experiencing at Least One Adverse Event (AE) During the Treatment Period and First 14 Follow-up Days
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol -specified procedure, whether or not considered related to the medicinal product or protocol -specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: 14 days following last dose of study drug (up to 26 weeks)
Population: All Participants as Treated (APaT) Population; all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 29 | 28 | 30
participants | 28 | 28 | 28

3. Primary Outcome: Number of Participants Discontinued From Study Treatment Due to AEs During the Treatment Period and First 14 Follow-up Days
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol -specified procedure, whether or not considered related to the medicinal product or protocol -specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to 24 weeks
Population: APaT Population; all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 29 | 28 | 30
participants | 1 | 1 | 1

4. Secondary Outcome: Percentage of Participants Achieving Undetectable HCV RNA During Treatment by Time Point
Description: HCV RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay on blood samples drawn from each participant at Week 2, Week 4, Week 12, and at end of treatment. The assay has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. Undetectable HCV RNA was defined as HCV RNA < 9.3 IU/mL.
Time Frame: From Treatment Week (TW) 2 through end of treatment (up to 24 weeks)
Population: Participants in the PP Population (all randomized participants receiving ≥1 dose of study treatment and no important protocol deviation) with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 29 | 26 | 29
percentage of participants
  Week 2 (n=29, 25, 29) | 34.5 [17.9 to 54.3] | 32.0 [14.9 to 53.5] | 55.2 [35.7 to 73.6]
  Week 4 (n=28, 26, 29) | 82.1 [63.1 to 93.9] | 76.9 [56.4 to 91.0] | 89.7 [72.6 to 97.8]
  Week 12 (n=28, 26, 28) | 96.4 [81.7 to 99.9] | 92.3 [74.9 to 99.1] | 100.0 [87.7 to 100.0]
  End of All Therapy (n=26, 25, 26) | 92.3 [74.9 to 99.1] | 92.0 [74.0 to 99.0] | 100.0 [86.8 to 100.0]

5. Secondary Outcome: Percentage of Participants Achieving HCV RNA <25 IU/mL During Treatment by Time Point
Description: HCV RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay on blood samples drawn from each participant at Week 2, Week 4, Week 12, and at end of treatment. The assay has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL.
Time Frame: From TW 2 through end of treatment (up to 24 weeks)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 29 | 26 | 29
percentage of participants
  Week 2 (n=29, 25, 29) | 86.2 [68.3 to 96.1] | 88.0 [68.8 to 97.5] | 96.6 [82.2 to 99.9]
  Week 4 (n=28, 26, 29) | 96.4 [81.7 to 99.9] | 100.0 [86.8 to 100.0] | 100.0 [88.1 to 100.0]
  Week 12 (n=28, 26, 28) | 96.4 [81.7 to 99.9] | 100.0 [86.8 to 100.0] | 100.0 [87.7 to 100.0]
  End of all Therapy (n=26, 25, 26) | 92.3 [74.9 to 99.1] | 100.0 [86.3 to 100.0] | 100.0 [86.8 to 100.0]

6. Secondary Outcome: Percentage of Participants Achieving SVR4
Description: HCV RNA was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. SVR4 was defined as HCV RNA <25 IU/mL (either target detected, unquantifiable or target not detected) 4 weeks after the end of all study therapy.
Time Frame: 4 weeks after end of treatment (up to 28 weeks total)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 26 | 25 | 26
percentage of participants | 76.9 [56.4 to 91.0] | 88.0 [68.8 to 97.5] | 92.3 [74.9 to 99.1]

7. Secondary Outcome: Percentage of Subjects Achieving SVR24
Description: HCV RNA was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. SVR24 was defined as HCV RNA <25 IU/mL (either target detected, unquantifiable or target not detected) 24 weeks after the end of all study therapy.
Time Frame: 24 weeks after end of treatment (up to 48 weeks total)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 24 | 25 | 26
percentage of participants | 54.2 [32.8 to 74.4] | 84.0 [63.9 to 95.5] | 84.6 [65.1 to 95.6]

8. Secondary Outcome: Number of Participants Developing Post-baseline Antiviral Resistance to Grazoprevir Among Participants Not Achieving SVR24 Response
Description: Post-baseline resistance associated variants (RAV) analysis was conducted by comparing the amino acid sequences at virologic failure time points to those at baseline (BL): Day 1, pre-dose. A post-BL variant was defined as an amino acid substitution within HCV NS3/4A that was present after the first dose at virologic failure and follow-up visits but not at BL. Post-BL variant analysis was conducted for participants who did not achieve SVR24 who had sequence data available.
Time Frame: From Day 1 up to Follow-up Week 24 (up to 48 weeks total)
Population: Treated non-SVR24 participants with BL and post-BL samples sequenced for RAVs.
Measure: Number; unit: participants
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Number analyzed (Participants) | 12 | 7 | 4
participants | 9 | 5 | 3

ADVERSE EVENTS:
Time Frame: From 1st day of treatment (Day 1) through Follow-up Week 24 (up to 48 weeks)
Description: AEs were reported for the APaT Population (all randomized participants who received at least one dose of study treatment) during the treatment period and entire follow-up period.
Arm/Group | Grazoprevir 25 mg + PEG-IFN + RBV | Grazoprevir 50 mg + PEG-IFN + RBV | Grazoprevir 100 mg + PEG-IFN + RBV
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/28 | 0/30
Other Adverse Events (participants affected / at risk) | 28/29 | 28/28 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 25 mg + PEG-IFN + RBV (N=29) | Grazoprevir 50 mg + PEG-IFN + RBV (N=28) | Grazoprevir 100 mg + PEG-IFN + RBV (N=30)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 25 mg + PEG-IFN + RBV (N=29) | Grazoprevir 50 mg + PEG-IFN + RBV (N=28) | Grazoprevir 100 mg + PEG-IFN + RBV (N=30)
Anaemia (Blood and lymphatic system disorders) | 8 (11) | 11 (11) | 11 (11)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 3 (5)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 4 (5) | 7 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (3) | 2 (3)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (8) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 17 (18) | 9 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (6)
Asthenia (General disorders) | 2 (2) | 2 (2) | 3 (3)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 13 (14) | 12 (12) | 13 (13)
Fatigue (General disorders) | 18 (18) | 17 (17) | 18 (19)
Feeling cold (General disorders) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 6 (6) | 7 (7) | 7 (7)
Injection site erythema (General disorders) | 9 (9) | 8 (8) | 7 (7)
Irritability (General disorders) | 8 (8) | 2 (2) | 7 (8)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Pain (General disorders) | 3 (5) | 2 (2) | 6 (6)
Pyrexia (General disorders) | 10 (12) | 7 (7) | 11 (11)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (6) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 3 (4)
Red cell distribution width increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 7 (7) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 6 (7) | 9 (10)
Disturbance in attention (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 5 (6) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 10 (13) | 17 (19) | 13 (17)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 4 (5)
Chromaturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (9) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.